CLINICAL TRIAL: NCT00157183
Title: Non-invasive Ventilation and Oxygen Therapy in Cystic Fibrosis Patients With Nocturnal Oxygen Desaturation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); Monash University (Other); Cystic Fibrosis Federation Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 35/03
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; hypoxia; oxygen; noninvasive ventilation; quality of life
MeSH Terms: conditions — Cystic Fibrosis; Hypoxia

INTERVENTIONS:
Device: Nocturnal oxygen , nocturnal bi-level positive pressure ventilation

SUMMARY:
The purpose of this study is to determine whether correction of low nighttime oxygen (O2) levels and/ or high carbon dioxide levels in patients with cystic fibrosis improves their quality of life. The treatments being used overnight are (1)O2 (2)pressurised air which assists breathing (non-invasive positive pressure ventilation, NIPPV)

DETAILED DESCRIPTION:
Cystic fibrosis is the commonest life-limiting genetic disorder in the Caucasian population with a median survival of 31 years. Lung disease is responsible for the majority of morbidity and mortality and correlates with declining quality of life. Respiratory failure is the primary cause of death. Daytime respiratory failure (hypoxia with pO2<55 and/or hypercapnia with pCO2>50) is associated with a worse prognosis with a 2-year survival of 50%. Nocturnal respiratory failure (greater than 5% of the night spent with SpO2<90% and/or rise in PtcCO2>10mmHg overnight) is a precursor to the development of daytime respiratory failure. It has been postulated that earlier treatment of respiratory failure may improve outcome and quality of life.

Intervention: Nocturnal O2 and bilevel NIPPV in CF patients with nocturnal respiratory failure, compared to nocturnal placebo (air). Crossover trial utilising patients as their own control.

Aims: (1) To assess the effects of non-invasive ventilation (NIV) and oxygen (O2) therapy on quality of life, hospital admission rate, sleep quality and exercise tolerance in CF patients with NRF (2) To identify a level of severity of NRF where treatment with NIV is effective

ELIGIBILITY:
Inclusion Criteria:

proven diagnosis cystic fibrosis, age 18 years or older, FEV1< 70% predicted normal, clinically stable (no admission or antibiotics last 2 weeks, OR end of admission where further clinical improvement not expected), nocturnal respiratory failure (SpO2<90% for > 10% of night or rise in PtcCO2 > 5 mmHg in REM), daytime hypercapnia (PaCO2> 45 mmHg)

Exclusion Criteria:

Previous home O2 or NIV use, Sedative medications, Cardiac/renal/endocrine/neurological disease likely to compromise ventilatory control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaires:
CFQoL questionnaire (Gee,Thorax,2000)(a priori chest, physical function, treatment, emotion domains)
Epworth Sleepiness Scale
Pittsburgh Sleep Quality Index
CF Subjective Symptoms Sleep disturbance Questionnaire (CSQ-in house)
Medical Research Council Dyspnea Scale
Baseline Dyspnea Index, Transitional Dyspnea Index
Work or Study status
Physiological:
Nocturnal SpO2, nocturnal rise in transcutaneous CO2
Daytime arterial blood gases (PaCO2, PaO2)

SECONDARY OUTCOMES:
Admission rate
Lung function tests (FEV1, FVC, RV/ TLC)
Modified CF shuttle walk test
Neurocognitive testing (psychomotor vigilance task, Stroop, Controlled Oral Word Association Test, Trails A and B, digit recall forwards backwards)
PSG (sleep efficiency, arousal index, % REM sleep, urinary catecholamines)
Serum cytokines (IL-6, TNF alpha, IL-1 beta)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Naughton, MD, Principal Investigator — The Alfred
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Young AC, Wilson JW, Kotsimbos TC, Naughton MT. The impact of nocturnal oxygen desaturation on quality of life in cystic fibrosis. J Cyst Fibros. 2011 Mar;10(2):100-6. doi: 10.1016/j.jcf.2010.11.001. Epub 2010 Dec 30. PMID 21195036